CLINICAL TRIAL: NCT00038480
Title: A Phase I/II Study of Lopinavir/Ritonavir in HIV-1 Infected Infants Less Than 6 Months of Age
Brief Title: Safety and Effectiveness of Lopinavir/Ritonavir in HIV Infected Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1030; 10041 (Registry Identifier: DAIDS ES); PACTG P1030
Record Dates: First submitted 2002-05-31; First posted 2002-06-03 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Lopinavir; HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir

INTERVENTIONS:
Drug: Lopinavir/Ritonavir

SUMMARY:
The purpose of this study is to find out if the drug lopinavir/ritonavir (LPV/RTV) is safe and well tolerated in HIV infected infants. This study will also determine the most effective dose of LPV/RTV for infants.

DETAILED DESCRIPTION:
LPV/RTV has shown significant antiviral activity and tolerability in clinical trials in adults and children over 6 months of age. LPV/RTV has been approved by the FDA to treat older children and adults with HIV. Data for children under 6 months, however, have not been available. LPV/RTV has not been approved for infants less than 6 months old, and the appropriate dose for young infants is not known. Dosing guidelines are needed for young infants, most of whom are in the early stages of primary infection. This study will help identify an appropriate dose range of LPV/RTV and evaluate response to therapy in infants less than 6 months of age. The study will also evaluate whether early therapy allows normal development of the immune system.

Infants between 14 days and 6 months of age will receive LPV/RTV in combination with 2 nucleoside reverse transcriptase inhibitors (NRTIs) chosen by their physicians. Twelve-hour pharmacokinetic sampling is performed on Day 14 of drug treatment and when the patient reaches 12 months of age. Patients will undergo a physical exam, medical history assessment, and blood collection at selected study visits. Study visits will occur every 2 weeks for the first 8 weeks, then every 4 weeks until the end of the first year of the study. Study visits during the second year will be every 12 weeks until the end of the study. The parent or guardian will be contacted by phone every 6 weeks to monitor adverse drug effects. Participants between the ages of 6 weeks but less than 6 months old will be followed for 96 weeks after the enrollment of the last participant. Participants between the ages of 14 weeks but less than 6 weeks will be followed for 48 weeks after the enrollment of the last participant.

ELIGIBILITY:
Inclusion Criteria

* HIV infected
* Viral load greater than 10,000 copies/ml within 30 days prior to study entry
* Weigh more than 5.5 lbs at the time of enrollment
* Agree to take 2 nucleoside reverse transcriptase inhibitors (NRTIs) in addition to LPV/RTV
* Have consent of parent or guardian willing to provide signed informed consent and to have the infant followed at a PACTG site

Exclusion Criteria

* Currently taking a nonnucleoside reverse transcriptase inhibitor or protease inhibitor (PI) while on study
* Previously used LPV/RTV. Patients who were treated previously with other PIs are not excluded. Prior or concurrent maternal treatment with LPV/RTV is not excluded.
* For patients less than 6 weeks old at time of enrollment, less than 34 weeks gestation at delivery OR for patients 6 or more weeks old at time of enrollment, less than 32 weeks gestation at delivery
* Any laboratory toxicity of Grade 3 or greater. Hyperlipasemia of Grade 2 or higher is also excluded.
* Newly diagnosed acute opportunistic or serious bacterial infection requiring therapy at the time of enrollment
* Chemotherapy for active cancer
* Certain medications
* Any other clinically significant conditions, other than HIV infection, that would interfere with the study

Ages: 14 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Trough concentration of LPV and pharmacokinetic parameters | Weeks 8, 16, 24, 36, 48, 60, 72, 84, and 96
Recurrent treatment-related Grade 3 and non-life threatening Grade 4 toxicity or single occurence of life-threatening Grade 4 toxicity | Throughout study

SECONDARY OUTCOMES:
Change in CD4 and CD8 count and percentage from baseline. HIV-1 specific CD4 count and CD8 mediated and humoral responses | Study entry and Weeks 12, 24, 36, 48, 60, 72, 84, and 96
Time to virologic failure | Throughout study
Suppression of viral load to less than 400 copies/ml and less than 50 copies/ml | Study entry and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 36, 40, 48, 60, 72, 84, and 96

CONTACTS AND LOCATIONS:
Overall Officials: Ellen G. Chadwick, MD, Study Chair — Children's Memorial Hospital, Division of Pediatric Infectious Diseases; Jorge Pinto, MD, DSc, Study Chair — Escola de Medicine, Universidade Federal de Minas Gerais
Locations (17):
- United States (14):
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Children's National Med. Ctr. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - USF - Tampa NICHD CRS, Tampa, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - St. Jude/UTHSC CRS, Memphis, Tennessee
- Brazil (2):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Minas Gerais
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Luzuriaga K, Wu H, McManus M, Britto P, Borkowsky W, Burchett S, Smith B, Mofenson L, Sullivan JL. Dynamics of human immunodeficiency virus type 1 replication in vertically infected infants. J Virol. 1999 Jan;73(1):362-7. doi: 10.1128/JVI.73.1.362-367.1999. PMID 9847340
- [Background] Equils O, Garratty E, Wei LS, Plaeger S, Tapia M, Deville J, Krogstad P, Sim MS, Nielsen K, Bryson YJ. Recovery of replication-competent virus from CD4 T cell reservoirs and change in coreceptor use in human immunodeficiency virus type 1-infected children responding to highly active antiretroviral therapy. J Infect Dis. 2000 Sep;182(3):751-7. doi: 10.1086/315758. Epub 2000 Aug 15. PMID 10950768
- [Background] Luzuriaga K, McManus M, Catalina M, Mayack S, Sharkey M, Stevenson M, Sullivan JL. Early therapy of vertical human immunodeficiency virus type 1 (HIV-1) infection: control of viral replication and absence of persistent HIV-1-specific immune responses. J Virol. 2000 Aug;74(15):6984-91. doi: 10.1128/jvi.74.15.6984-6991.2000. PMID 10888637
- [Background] Saez-Llorens X, Violari A, Deetz CO, Rode RA, Gomez P, Handelsman E, Pelton S, Ramilo O, Cahn P, Chadwick E, Allen U, Arpadi S, Castrejon MM, Heuser RS, Kempf DJ, Bertz RJ, Hsu AF, Bernstein B, Renz CL, Sun E. Forty-eight-week evaluation of lopinavir/ritonavir, a new protease inhibitor, in human immunodeficiency virus-infected children. Pediatr Infect Dis J. 2003 Mar;22(3):216-24. doi: 10.1097/01.inf.0000055061.97567.34. PMID 12634581
- [Result] Chadwick EG, Pinto J, Yogev R, Alvero CG, Hughes MD, Palumbo P, Robbins B, Hazra R, Serchuck L, Heckman BE, Purdue L, Browning R, Luzuriaga K, Rodman J, Capparelli E; International Maternal Pediatric Adolescent Clinical Trials Group (IMPAACT) P1030 Team. Early initiation of lopinavir/ritonavir in infants less than 6 weeks of age: pharmacokinetics and 24-week safety and efficacy. Pediatr Infect Dis J. 2009 Mar;28(3):215-9. doi: 10.1097/INF.0b013e31818cc053. PMID 19209098
- [Result] Chadwick EG, Yogev R, Alvero CG, Hughes MD, Hazra R, Pinto JA, Robbins BL, Heckman BE, Palumbo PE, Capparelli EV; International Pediatric Adolescent Clinical Trials Group (IMPAACT) P1030 Team. Long-term outcomes for HIV-infected infants less than 6 months of age at initiation of lopinavir/ritonavir combination antiretroviral therapy. AIDS. 2011 Mar 13;25(5):643-9. doi: 10.1097/QAD.0b013e32834403f6. PMID 21297419
- [Derived] Persaud D, Palumbo PE, Ziemniak C, Hughes MD, Alvero CG, Luzuriaga K, Yogev R, Capparelli EV, Chadwick EG. Dynamics of the resting CD4(+) T-cell latent HIV reservoir in infants initiating HAART less than 6 months of age. AIDS. 2012 Jul 31;26(12):1483-90. doi: 10.1097/QAD.0b013e3283553638. PMID 22555165
- [Derived] Persaud D, Palumbo P, Ziemniak C, Chen J, Ray SC, Hughes M, Havens P, Purswani M, Gaur AH, Chadwick EG; Pediatric AIDS Clinical Trials Group P1030 Team. Early archiving and predominance of nonnucleoside reverse transcriptase inhibitor-resistant HIV-1 among recently infected infants born in the United States. J Infect Dis. 2007 May 15;195(10):1402-10. doi: 10.1086/513871. Epub 2007 Apr 5. PMID 17436219